CLINICAL TRIAL: NCT00415181
Title: The Pharmacogenomics of Paclitaxel in Patients With Ovarian Cancer: Predictors of Toxicity and Response
Brief Title: Pharmacogenomics of Paclitaxel in Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Danish Clinical Intervention Research Academy (Other); Ministry of the Interior and Health, Denmark (Other Government)
Responsible Party: Troels K Bergmann, University of Southern Denmark
Other Study IDs: AKF-319pro
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2006-12

CONDITIONS: Ovarian Neoplasms; Fallopian Tube Neoplasms
Keywords: CYP2C8; MDR1; Pharmacogenetics; Paclitaxel
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood

SUMMARY:
This study will try to determine whether or not certain genes are responsible for the huge variation in toxicity and effect observed between patients treated with paclitaxel (chemotherapeutic drug). Specifically we will study this in patients with ovarian cancer who receive paclitaxel/carboplatin chemotherapy after primary surgery.

DETAILED DESCRIPTION:
Paclitaxel is an antineoplastic drug used in the treatment of ovarian cancer. The effect and toxicity is unpredictable in the individual patient. Paclitaxel is removed (eliminated) from the organism by oxidation. CYP2C8 is the enzyme mainly responsible. P-glycoprotein (Pgp) is an efflux transport protein natural to the human organism. Pgp is responsible for excretion of drugs via the bile and the kidneys and is thought to play a role in chemotherapy resistance. Paclitaxel is substrate for Pgp. Single nucleotide polymorphisms are possible causes for variation in both CYP2C8 and Pgp expression/function. We will study a possible role of these genetic variations as predictors of paclitaxel toxicity and effect and the possible implications for individual dosing in the future.

We want to determine the metabolic capacity of approximately 100 ovarian cancer patients and comparing this with genotypes, acute toxicity(eg. bone marrow suppression and neuropathy) and response to treatment(ie. CA125 response, progression free survival and overall survival). The metabolic capacity is estimated using a "sparse sampling" approach applying advanced computerized pharmacokinetic/dynamic modelling as opposed to traditional "frequent sampling" pharmacokinetic studies which burden the individual patient more.

Patients are recruited in collaboration with Oncological departments throughout Scandinavia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnose and histology of invasive epithelial ovarian/tuba or peritoneal cancer
* FIGO stage IIb-IV any grade or FIGO Ia-IIa only grade 3 or clear cell carcinoma (any stage and grade)
* Natural candidate for paclitaxel 175mg/m2 + Carboplatin (AUC=5-6)
* Baseline CA125≥70 AND/OR evaluable disease after RECIST (incl ultrasound)
* 18 years or older
* Caucasian (ie.parents and grandparents are Caucasian)
* Performance status 2 or lower (after WHO/ECOG)

Exclusion Criteria:

* Prior malignant disease apart from cervical carcinoma in situ and basal cell carcinoma of the skin
* Prior chemo / radiotherapy
* Ongoing or imminent other chemotherapies
* Pregnant or lactating
* Fertile woman of childbearing potential not willing to use adequate contraception
* Neurological symptoms (any kind) worse than CTCAE grade 1
* Active infection or other serious disease that could impair on treatment and/or follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2006-09; Primary Completion 2009-01 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Brøsen, phd, Study Director — University of Southern Denmark
Locations (4):
- Denmark (3):
  - Department of oncology, Herlev Hospital, Herlev
  - Department of Oncology, Odense University Hospital, Odense
  - Department of Oncology, Vejle Hospital, Vejle
- Department of Oncology, University Hospital of Lund, Lund, Sweden

REFERENCES:
- [Result] Bergmann TK, Brasch-Andersen C, Green H, Mirza M, Pedersen RS, Nielsen F, Skougaard K, Wihl J, Keldsen N, Damkier P, Friberg LE, Peterson C, Vach W, Karlsson MO, Brosen K. Impact of CYP2C8*3 on paclitaxel clearance: a population pharmacokinetic and pharmacogenomic study in 93 patients with ovarian cancer. Pharmacogenomics J. 2011 Apr;11(2):113-20. doi: 10.1038/tpj.2010.19. Epub 2010 Apr 6. PMID 20368717